CLINICAL TRIAL: NCT06768268
Title: Advanced Research on ICG Fluorescence Imaging-Guided Surgery Technique Using Mannitol and Voluven as Adjuncts
Brief Title: A Dose-Image Optimization Trial Evaluating Mannitol and Voluven as Adjuncts for Indocyanine Green
Acronym: ICGMV
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Yang Ming Chiao Tung University (Other); National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 202409024MIND; 114-BIH052 (Other Grant/Funding Number: National Taiwan University Hospital Hsinchu Branch)
Record Dates: First submitted 2024-12-29; First posted 2025-01-10 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: indocyanine green; sentinel lymph node biopsy; near-infrared fluorescence; 6-hydroxyethyl starch; mannitol; breast cancer; fluorescence-guided surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Mannitol

STUDY DESIGN:
Intervention Model Description: The study is a dose-escalation trial of adding Mannitol into Voluven-ICG solution as solvent/adjunct. The patients will be invited in groups of three, and the proportion of Mannitol will be escalated in the sequential groups.
Who Masked: Participant
Masking Description: The participants will not know which concentration group they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Pure Voluven (Active Comparator): The solution is prepared using Voluven as solvent, forming a 0.25 mg/mL ICG:Voluven solution.
  Interventions: Procedure: Voluven-assisted Indocyanine green fluorescence guided sentinel lymph node biopsy for breast cancer
- 1:10 (Active Comparator): The solution is prepared using Mannitol(20%):Voluven=1:10 as solvent, forming a 0.25 mg/mL ICG:Solvent solution.
  Interventions: Procedure: Voluven-assisted Indocyanine green fluorescence guided sentinel lymph node biopsy for breast cancer; Drug: Mannitol (20%)
- 1:8 (Active Comparator): The solution is prepared using Mannitol(20%):Voluven=1:8 as solvent, forming a 0.25 mg/mL ICG:Solvent solution.
  Interventions: Procedure: Voluven-assisted Indocyanine green fluorescence guided sentinel lymph node biopsy for breast cancer; Drug: Mannitol (20%)
- 1:6 (Active Comparator): The solution is prepared using Mannitol(20%):Voluven=1:6 as solvent, forming a 0.25 mg/mL ICG:Solvent solution.
  Interventions: Procedure: Voluven-assisted Indocyanine green fluorescence guided sentinel lymph node biopsy for breast cancer; Drug: Mannitol (20%)
- 1:4 (Active Comparator): The solution is prepared using Mannitol(20%):Voluven=1:4 as solvent, forming a 0.25 mg/mL ICG:Solvent solution.
  Interventions: Procedure: Voluven-assisted Indocyanine green fluorescence guided sentinel lymph node biopsy for breast cancer; Drug: Mannitol (20%)

INTERVENTIONS:
Procedure: Voluven-assisted Indocyanine green fluorescence guided sentinel lymph node biopsy for breast cancer — The procedure includes: (1) preparation of specific formula of ICG:Voluven solution (2) injection of ICG solution at subarelar area or peri-tumoral area (3) observation of fluorescent lymphatic drainage and retrieval of sentinel lymph nodes
Drug: Mannitol (20%) — Adding Mannitol into Voluven and used as solvent of ICG
  Arms: 1:10; 1:4; 1:6; 1:8

SUMMARY:
The goal of this clinical trial is to exploring the use of Mannitol 20% as a solvent to prepare ICG solution, combining with Voluven, forming a hybrid small-large molecular weight solvent for protecting ICG in monomer form and stimulating lymphatic uptake simultaneously in early breast cancer patients who is indicated to undergo sentinel lymph node biopsy. The main question it aims to answer is:

* Will adding Mannitol with Voluven as ICG solvent improve the fluorescence signal of the lymph nodes, comparing with using pure Voluven?
* Which proportion of Mannitol-Voluven delivers the best image quality when used as solvent of ICG?

Researchers will compare the following arms with different solvent (all arms' final ICG concentration are 0.25mg/mL):

* Pure Voluven
* Mannitol:Voluven = 1:10
* Mannitol:Voluven = 1:8
* Mannitol:Voluven = 1:6
* Mannitol:Voluven = 1:4 to see if increased Mannitol:Voluven ratio as ICG solvent translates to better fluorescence image quality.

Participants will be invited in a group of 3, and be blindly assigned to each concentration group sequentially. Participants will undergo ICG fluorescence guided sentinel lymph node biopsy with the assigned solution formula. The endpoints included number of lymph nodes obtained, fluorescence signal-to-background ratio of the lymph nodes, lymphatic uptake rate, lymphatic drainage speed, detection method, lymph node pathology, and any intra- or post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult females aged 20 to 70 years old.
* Pathologically confirmed invasive breast cancer patients who are eligible for sentinel lymph node biopsy.

Exclusion Criteria:

* History of allergy to iodine, ICG, blue dye, Voluven, or Mannitol.
* History of hyperthyroidism, thyroid cancer, etc.
* Current pregnancy, lactation, or breast infection.
* Individuals with impaired mental capacity or belonging to vulnerable populations.
* Patients who have undergone neoadjuvant chemotherapy prior to surgery.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of sentinel lymph nodes | From the procedure day to the follow-up clinic visit day (average 10 days)
  The number of the retrieved sentinel lymph nodes
Fluorescence signal-to-background ratio of the lymph nodes | From the procedure day to the follow-up clinic visit day (average 10 days)

SECONDARY OUTCOMES:
Lymphatic uptake rate | From the procedure day to the follow-up clinic visit day (average 10 days)
  The time from injection to the development of fluorescent subcutaneous lymphatics
Lymphatic drainage speed | From the procedure day to the follow-up clinic visit day (average 10 days)
  The time from the initiation of visible fluorescent subcutaneous lymphatics to that reaches the axilla
Detection method | From the procedure day to the follow-up clinic visit day (average 10 days)
  The method of the sentinel lymph node being detected. (Could be radioisotope, blye dye, ICG fluorescence, or combination of multiple methods)
Lymph node pathology | From the procedure day to the follow-up clinic visit day (average 10 days)
  The positivity of sentinel lymph node metastasis in the pathology report.

CONTACTS AND LOCATIONS:
Overall Officials: Yung Chun Hsieh, M.D., MMSC, Study Chair — National Taiwan University Hospital Hsinchu Branch
Locations (1):
- National Taiwan University Hospital Hsinchu Branch, Hsinchu County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hsieh YC, Guo KW, Wang MW, Su SP, Syu YH, Huang CS, Chan YH. A Novel Injection Protocol Using Voluven(R)-Assisted Indocyanine Green with Improved Near-Infrared Fluorescence Guidance in Breast Cancer Sentinel Lymph Node Mapping-A Translational Study. Ann Surg Oncol. 2023 Dec;30(13):8419-8427. doi: 10.1245/s10434-023-14129-4. Epub 2023 Aug 21. PMID 37605084